CLINICAL TRIAL: NCT01770444
Title: Safety and Efficacy of Implementing Low-Dose Coronary Computed Tomographic Angiography for Early Triage of Acute Chest Pain in Emergency Department
Brief Title: Low-Dose Coronary Computed Tomographic Angiography for Early Triage of Acute Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: B-1211/177-005
Record Dates: First submitted 2012-12-20; First posted 2013-01-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2015-11

CONDITIONS: Chest Pain
Keywords: Acute coronary syndrome; Cardiac computed tomographic angiography; Radiation dose reduction; Medical radiation exposure
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose cardiac CT (Experimental): Patients randomized to this group will be assessed by low-dose cardiac CT protocol.
  Interventions: Other: Low-dose Cardiac CT protocol
- Conventional cardiac CT (Other): Patients randomized to this group will be assessed by conventional cardiac CT protocol.
  Interventions: Other: Conventional cardiac CT protocol

INTERVENTIONS:
Other: Low-dose Cardiac CT protocol — A cardiac CT protocol modified for reduction of radiation exposure
  1. Prospective gating
  2. Range: dedicated imaging (below carina to heart base)
  Arms: Low-dose cardiac CT
Other: Conventional cardiac CT protocol — Conventional CCTA protocol
  1. Retrospective gating with tube current modulation
  2. Range: dedicated imaging (below carina to heart base)
  Arms: Conventional cardiac CT

SUMMARY:
This study is to see whether the low-dose coronary computed tomographic angiography (CCTA) protocol is as safe and efficacious as conventional-dose protocol in early triage of acute chest pain.

DETAILED DESCRIPTION:
Currently, CCTA is a valuable tool for early triage of low to intermediate risk acute chest pain patients in emergency department. However, it has been criticized for causing unnecessary radiation exposure in the population where its majority has no coronary lesion. A low-dose CCTA protocol comprised with 1) dedicated cardiac imaging protocol (rather than triple rule-out protocol), 2) prospective gating and 3) without additional imaging for calcium scoring will be used to implement the low-dose imaging. We hypothesized that the low-dose CCTA protocol will be as safe and efficacious as conventional dose protocol while decreasing the amount of radiation exposure significantly.

ELIGIBILITY:
Inclusion Criteria:

- Patients visiting emergency department for A) acute onset (<12hr) chest pain or equivalent symptoms B) aged between 25-55, C) that requires to rule out acute coronary syndrome.

Exclusion Criteria:

1. Known coronary artery disease and/or any related intervention (STENT, CABG)
2. Elevated cardiac biomarkers (CK-MB, Troponin I)
3. Ischemic ECG changes
4. Documented evidence of low LV systolic function (ejection fraction ≤ 45%)
5. TIMI risk >4
6. Unstable vital sign (e.g. hypoxemia, shock)
7. Patients with contraindication to iodinated contrast and/or beta blockers including renal failure or reactive airway diseases such as COPD or asthma
8. Atrial fibrillation on initial ECGs
9. Active renal disease, serum creatinine ≥1.5 mg/dl
10. Negative coronary angiography or CCTA within 6 months
11. Modified Wells criteria >4 or D-dimer > 0.5ug/mL
12. Suspicious of aortic dissection or D-dimer > 0.5ug/mL

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 681 (Actual)
Dates: Start 2012-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having hard events (death, MI) after negative low-dose CCTA findings | Within one month after discharge from emergency department

SECONDARY OUTCOMES:
Direct comparison of accuracy (sensitivity, specificity, PPV, NPV) for between low-dose and conventional cardiac CT | One month after discharge from emergency department
  The diagnostic accuracy of detecting ACS will be assessed using patient chart review and telephone interview (48-72 hours and one month after discharge) as appropriate. ACS event (and MACE) will be adjudicated by independent cardiologists.
Direct comparison of frequency and overall cost of additional tests such as echocardiography, treadmill test, myocardial SPECT and coronary angiography | During 1) index ED visit, which will be an average of 1 day and 2) one-month follow-up period after discharge
Total radiation dose exposed by index CT imaging and additional tests including SPECT and invasive angiography | During 1) index ED visit, which will be an average of 1 day and 2) one-month follow-up period after discharge
Total length of ED and hospital stay | Time spent for index ED visit, which will be an average of 24 hours and total hospital stay until discharge, which will be an average of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuseok Kim, MD, Study Director — Department of emergency medicine, Seoul national university Bundang hospital; Sangil Choi, MD, Study Director — Department of radiology, Seoul national university Bundang hospital
Locations (3):
- South Korea (3):
  - Seoul national university Bundang hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Seoul national university Boramae medical center, Seoul